## THE EFFECT OF EDUCATION GIVEN BEFORE PORT CATHETER INFUSION ON INFUSION RELATED SYMPTOMS

Yekta DEMİRSOY

## **EVALUATION OF DATA**

The data obtained in the study will be analyzed using the SPSS (Statistical Package for Social Sciences) for Windows 22.0 program. The Kolmogorov Smirnov Test will be used to determine whether the research data is normally distributed. According to the Kolmogorov Smirnov Test, if p>0.05, the distribution is determined to be normal.

However, if p<0.05, the distribution is determined to be non-normal and the Skewness and Kurtosis values of the data are examined. If the Skewness and Kurtosis values are between +2 and -2, the variable is considered to be normally distributed. The homogeneity of the descriptive characteristics between the groups will be tested with chi-square analysis. For the difference between the means of two independent groups, if the data is normally distributed, the t-test will be used, and if the data is not normally distributed, the Mann-Whitney U test will be used. Changes in measurements within the group will be analyzed with the repeated measures Anova test if the data is normally distributed, and if the data is not normally distributed, the Friedman test will be used.

## IMPLEMENTATION OF THE STUDY

The rationale and purpose of the study will be explained to patients who meet the inclusion criteria. Written informed consent will be obtained from patients who agree to participate in the study. Patients will be assigned to the intervention and control groups with simple randomization. Patients in both groups will be administered the Patient Identification Form and State-Trait Anxiety Scale before the port catheter needle insertion procedure. Blood pressure, heart rate, respiratory rate, oxygen saturation, urination-related anxiety and visual analog scale will be measured and recorded in the Symptom Chart

(Pre-test). Patients in the experimental group will be informed by the researcher about the educational content created regarding the port catheter needle insertion procedure and breathing exercises. The researcher will watch the educational content and answer the questions of the experimental group patients. No educational content will be administered to the control group patients. Port catheter needle insertion will be applied to both groups. After the procedure is completed, the State and Trait Anxiety Scale and the Symptom Schedule from the data collection tools will be re-applied to the patients in both groups (Post-test).